CLINICAL TRIAL: NCT03241186
Title: Single Arm Phase II Study of Ipilimumab and Nivolumab as Adjuvant Therapy for Resected Mucosal Melanoma (SALVO Study). HCRN: MEL16-252
Brief Title: Ipilimumab and Nivolumab as Adjuvant Treatment of Mucosal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Robert R. McWilliams, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Robert R. McWilliams, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEL16-252
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Mucosal Melanoma
Keywords: Ipilimumab; Nivolumab; OPDIVO; IgG4 kappa immunoglobulin
MeSH Terms: interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ipilimumab (1 mg/kg) + Nivolumab (3 mg/kg) IV (Experimental): Cycles 1-4: Ipilimumab (1 mg/kg) + Nivolumab (3 mg/kg) IV Day 1 of each Cycle Each Cycle = 21 days
  Cycles 5-15: Nivolumab IV 480 mg Day 1 of each Cycle Each Cycle = 28 days
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — 1mg/kg
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Nivolumab — 3mg/kg
  Other Names: OPDIVO; BMS-936558; ONO-4538; MDX1106
Drug: Nivolumab — 480mg
  Other Names: OPDIVO; BMS-936558; ONO-4538; MDX1106

SUMMARY:
This is a single arm phase II clinical trial of Ipilimumab and Nivolumab in patients with resected mucosal melanoma. Ipilimumab (1 mg/kg) and Nivolumab (3 mg/kg) will be administered Day 1 of a 21-day cycle in Cycles 1-4 and then nivolumab 480 mg will be administered Day 1 of a 28-day cycle for Cycles 5-15 (maximum of 15) or until disease recurrence or intolerance before completion of 15 cycles.

DETAILED DESCRIPTION:
Ipilimumab and Nivolumab Combination Administration

* Ipilimumab 1mg/kg given IV Day 1 for 3 weeks (21 days), for 4 cycles
* Nivolumab 3mg/kg given IV Day 1 for 3 weeks (21 days), for 4 cycles

Nivolumab Alone Administration

* Nivolumab 480mg given IV Day 1 for 4 weeks (28 days), for 5-15 cycles

Nivolumab is to be administered as an approximately 30-minute IV infusion (± 10 minutes). At the end of the infusion, flush the line with a sufficient quantity of normal saline.

Ipilimumab is to be administered as an approximately 30-minute IV infusion (± 10 minutes). At the end of the infusion, flush the line with a sufficient quantity of normal saline or 5% dextrose solution.

When both study drugs are to be administered on the same day, separate infusion bags and filters must be used for each infusion. Nivolumab is to be administered first. The nivolumab infusion must be promptly followed by a saline flush to clear the line of nivolumab before starting the ipilimumab infusion. The second infusion will always be ipilimumab, and will start at least 30 minutes after completion of the nivolumab infusion.

The dosing calculations should be based on the body weight from Cycle 1 Day 1. If the subject's weight on the day of dosing differs by > 5% from the weight used to calculate the dose, the dose should be recalculated based on the current day of treatment weight. All doses should be rounded to the nearest milligram. There will be no dose modifications allowed.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Histological confirmation of melanoma of any mucosal site including (but not limited to) anus/rectum, vulvar/vaginal, sinonasal. NOTE: Melanomas of cutaneous origin and/or ocular origin are ineligible.
* R0 or R1 resection of primary melanoma tumor (no gross disease can be left behind, but microscopically positive margins are acceptable).
* Surgery within ≤ 90 days of registration.
* ECOG Performance Status (PS) ≤ 1

The following laboratory values obtained ≤ 14 days prior to registration:

Hematological:

* Absolute Neutrophil Count (ANC) ≥ 1500/mm^3
* Hemoglobin (Hgb) ≥ 9 g/dL (may be transfused)
* Platelet (Plt) 100,000/mm^3

Renal:

* Serum Creatinine ≤ 1.5 x ULN

Hepatic:

* Alkaline Phosphatase (Alk Phos) ≤ 1.5 x upper limit of normal (ULN)
* Total and Direct Bilirubin ≤ 1.5 × (ULN)
* Aspartate aminotransferase (AST) ≤ 1.5 × ULN
* Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Willing to return to enrolling institution for follow-up
* Willing to provide archival tissue prior to C1D1 if available and blood samples for correlative research purposes

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the subject inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and subjects known to be HIV positive and currently receiving antiretroviral therapy. NOTE: Subjects known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* Other active malignancy ≤ 3 years prior to registration. EXCEPTIONS: Malignancies with a very low (< 5%) risk of recurrence such as non-melanotic skin cancer or carcinoma-in-situ of the cervix.
* History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.
* Active autoimmune disease -including but not limited to:

  * Subjects with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease,
  * Subjects with a history of symptomatic autoimmune disease requiring systemic treatment within the past 2 years with the use of disease modifying agents, corticosteroids, or immunosuppressive drugs.

    * rheumatoid arthritis
    * systemic progressive sclerosis (scleroderma)
    * systemic lupus erythematosus
    * psoriasis
    * autoimmune vasculitis (e.g., Wegener's Granulomatosis)
    * CNS or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome and Myasthenia Gravis, multiple sclerosis)

EXCEPTION: autoimmune conditions that are only requiring replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

* Any radiation within 2 weeks prior to study initiation. Neoadjuvant and adjuvant radiation are allowed, but must be completed > 2 weeks prior to registration.
* Any prior systemic therapy for melanoma (chemotherapy, immunotherapy, targeted therapy)
* Women of childbearing potential (WOCBP) must be willing to abstain from heterosexual intercourse or to use 2 forms of effective methods of contraception from the time of informed consent until 5 months after the last dose of study drug. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Examples include: intrauterine device (IUD), vasectomy of a female subject's male partner, contraceptive rod implanted into the skin, or use of two of the following: diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide), cervical cap with spermicide (nulliparous women only), contraceptive sponge (nulliparous women only), male condom or female condom (cannot be used together), hormonal contraceptive.*Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. NOTE: Male subjects are not required to utilize contraception. The study regimen is not genotoxic and systemic concentrations sufficient to produce a risk of fetal toxicity are not expected in WOCBP partners from exposure to a male participant's seminal fluid.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Assess Recurrence-free survival time (RFS) | 1.5 years
  Date the patient receives the first dose of study medication to the date of documentation of first disease recurrence or death due to any cause.

SECONDARY OUTCOMES:
Assess the Adverse Events | 2 years
  Adverse events will be graded and attribution assigned using CTCAE version 4
Overall Survival (OS) | 2 years
  The time from registration to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Robert R. McWilliams, MD, Study Chair — Hoosier Cancer Research Network
Locations (7):
- United States (7):
  - Mayo Clinic- Florida, Jacksonville, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org